CLINICAL TRIAL: NCT06471985
Title: CoPainHell: The Analgesic Effect of Alcohol and Music
Acronym: CPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eske Kvanner Aasvang (Other)
Responsible Party: Sponsor-Investigator, Eske Kvanner Aasvang, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CPH_2024
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Enya + Pain test (Active Comparator): In this arm, participants will listen to Enya in headphones while being exposed to the Cold Pressor Test.
  Interventions: Combination Product: Music and pain
- Slayer + Pain test (Active Comparator): In this arm, participants will listen to Slayer in headphones while being exposed to the Cold Pressor Test.
  Interventions: Combination Product: Music and pain

INTERVENTIONS:
Combination Product: Music and pain — In both arms of the study the participant will take the same pain test. They will either listen to Enya or slayer, depending on the arm

SUMMARY:
The study is a 2x2 randomized crossover study. Participants are randomized to listen to one of two music tracks: "Orinoco Flow" by Enya or "Raining Blood" by Slayer. Prior to the intervention, participants' breath alcohol levels are measured through a breathalyzer test. The intervention involves a cold water test, where the participant's dominant hand is submerged in water at 4-5 degrees Celsius. Participants are instructed to keep their hand in the water until the pain becomes too intense, but no longer than 5 minutes.

Two hours after the first test, the same procedure is repeated, but participants listen to the other music track than they did during the first test. Participants receive no instructions on how to behave during the 2-hour interval.

The experiment takes place during the music festival CopenHell (June 19-22, 2024), provided that there is approval from relevant authorities.

Two hours after the first test, the same procedure is repeated, but participants listen to the other music track than in the first test. Participants are given no instructions on how to behave during the 2-hour interval.

DETAILED DESCRIPTION:
This study is a 2x2 factorial randomized cross-over study investigating the effect of alcohol and music on analgesia. Enrollment will be at the Festival Site of Copenhell, Refshalevej 185, 1432 København K, Denmark. Participants meeting inclusion criteria will be enrolled.

Following the written and oral informed consent to participate in the trial, participants will fill out a questionnaire of demographics information.

When performing the intervention, participants will initially have their blood alcohol content measured with a breath analyzer measuring Breath Alcohol Content (BrAC). After BrAC measurement, the study participants will undergo ''cold pressor test'' (CPT) pain stimulation on their dominant arm:

Prior to the CPT, the participants will be randomized to either listening to the calm and relaxing song "Orinoco Flow" by Enya or the song "Raining Blood" by Slayer, considered one of the most iconic heavy-metal music numbers, during the test.

After the pain stimulation test the participants will undergo a wash out period lasting at least 2 hours where participants enjoy the festival on their own without any instructions.

Following the wash-out period the participants will return to another BrAC measurement followed by an identical CPT. However, this time they will listen to the opposite song than before. The investigators will expect that the participants will have a different alcohol concentration in the breath (higher/lower) for the second pain test.

The investigators will include up to 45 participants.

Explanation of Cold Pressor Test:

The CPT is performed with a cold-water bath with a temperature of 4° - 5° degrees cold circulating water. The participant will be asked to submerge their dominant hand and wrist in the cold water and a timer will be started simultaneously. Participants are asked to keep the hand in the water until pain threshold and pain tolerance is reached. Participants are allowed to move the hand or keep it still as they wish, and they are informed that there will be a time cap of 5 minutes to ensure no permanent damage.

The water will be circulated with an Eheim 1046 universal pump (Eheim, Deizisau, Germany), and temperature monitored with a Testo 925 waterproof precision thermometer (Testo, Lenzkirch, Germany). The CPT setup is identical to a prior study performed by the same author.

Prior to stimulation the participants will be thoroughly informed of the procedure by an investigator using the instructions of a previous study.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years old
* Informed consent
* Breath alcohol concentration ranging from 0.0 to 1.5 permille and deemed fit by the investigator at the time of giving informed consent

Exclusion Criteria:

* Wounds on dominant arm
* Current illness (a flu, cold etc.)
* Persons with diabetes because of the risk of peripheral neuropathies or other know peripheral sensibility paresthesia
* Circulation issues (especially Raynaud's syndrome)
* Pregnancy

Pull-out criteria

- Breath alcohol concentration > 2.5 permille and/or deemed unfit to participate by the investigator at the second pain test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
pain responsiveness | 300 seconds
  Pain responsiveness will be measured on the VAS, where an investigator will ask the participants to rate their experienced pain from 1-10.
  The VAS will be rated at the start of CPT + 30 seconds, 60 seconds, 90, 120, 180, 240 and 300 seconds or when reaching the pain tolerance (up to 5 minutes), where the test will end whichever comes first.
  VAS: Visuel Analog Scale. Values 0-10, where 0 is no pain at al and 10 is the worst pain imaginable

SECONDARY OUTCOMES:
pain threshold and pain tolerance | five minutes
  Pain threshold is measured as the number of seconds passed from the beginning of the pain stimulation till the participant says "pain", when stimulus evolves from being unpleasant to painful.
  Pain tolerance is measured as the number of seconds passed from the beginning of pain stimulation till the participant can't bear the pain anymore and says "pain limit".

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhell metal Festival, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No